CLINICAL TRIAL: NCT00575419
Title: Dose Escalation Study Of I.V. And Intra-Aortic N-Acetylcysteine For The Prevention Of Contrast Induced Nephropathy In Patients With Stage 3 Renal Failure Undergoing Contrast Imaging Studies: A Phase I Trial
Brief Title: Safety Study Of N-Acetylcysteine For Prevention Of Contrast Induced Nephropathy In Patients w/Stage 3 Renal Failure
Acronym: CIN-NAC
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Edward Neuwelt, Professor, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: OHSU-3673
Record Dates: First submitted 2007-12-14; First posted 2007-12-18 (Estimated); Last update posted 2019-08-02 (Actual); Status verified 2019-07

CONDITIONS: Contrast Induced Nephropathy
Keywords: Contrast Induced Nephropathy
MeSH Terms: interventions — Acetylcysteine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1, IV NAC (Experimental): N-acetylcysteine administered intravenously
  Interventions: Drug: N-acetylcysteine
- 2, IA NAC (Experimental): N-acetylcysteine administered intra-arterial
  Interventions: Drug: N-acetylcysteine

INTERVENTIONS:
Drug: N-acetylcysteine — * Dose Level 1: 150 mg/kg/day
  * Dose Level 2: 300 mg/kg/day
  * Dose Level 3: 600 mg/kg/day
  * Dose Level 4: 900 mg/kg/day
  * Dose Level 5: 1200 mg/kg/day

SUMMARY:
This will be a randomized prospective dose escalation clinical study of N-acetylcysteine (NAC) in patients with stage 3 or worse renal failure (Glomerular Filtration Rate 30-60 ml/min calculated with the Modification of Diet in Renal Disease formula), undergoing a procedure or imaging that requires the administration of contrast media at Oregon Health & Science University or the Portland Veterans Hospital. Subjects will receive NAC 60 minutes prior to the procedure or imaging requiring contrast media. Toxicity will be graded according to NCI Common Toxicity Criteria (CTC) version 3.0. An adult Phase 1 dose escalation study of NAC administered intravenously (IV) and intra-arterially (IA) will be performed. An isotonic nonionic contrast agent will be used in all cases. Contrast Induced Nephropathy (CIN) is defined as an increase in serum creatinine concentration of 25% or more from the subjects baseline value within a 72-hour period after the administration of contrast media. Serum creatinine concentration will be measured at admission, every day during in-patient hospitalization, and at hospital discharge.

DETAILED DESCRIPTION:
Radiographic contrast media is being used at an increasing rate for various diagnostic and therapeutic procedures. Renal failure following contrast administration for enhanced imaging has become a serious complication. Patients with underlying renal disorders have an increased incidence of Contrast Induced Nephropathy (CIN). CIN has been reported as the third most common cause of in-hospital renal failure after hypovolemia and post surgical renal insufficiency. Several factors increase the risk of CIN: preexisting renal dysfunction, volume and type of contrast agent employed, and lack of renal prophylaxis. CIN pathogenesis may be due to an injury to the renal cortex and outer medulla resulting from a decrease in blood flow, an osmotic effect, and/or direct toxicity to tubular cells by oxygen free radicals. N-acetylcysteine (NAC) is a cysteine analog and sulfur-containing agent, with strong antioxidant activity, which induces de novo synthesis of glutathione. NAC protection during the evolution of renal failure may be related to the ability to scavenge oxygen free radicals and/or improve endothelium-dependant vasodilation. There is no animal model that directly correlates with CIN, but the investigators have investigated nephrotoxicity and chemoprotection against cisplatin induced nephropathy which has a mechanism of action mediated through the generation of reactive intermediates in an animal model. NAC is potentially protective against cisplatin induced nephrotoxicity when administered at high intravenous (IV) doses (400 mg/kg) and at low intra-arterial (IA) doses (50mg/kg) down the descending aorta. This implies a safe dose-dependent effect of IV NAC and that lower doses can be used IA safely.

Objectives:

Primary Objective:

The primary objective of this study is to establish a maximum tolerated dose of both IV and IA NAC. This maximum tolerated dose will be evaluated primarily for efficacy in a future study.

Secondary Objectives:

1. To obtain data on changes from baseline serum creatinine and calculated creatinine clearance to provide sample size estimates for future studies.
2. To estimate the efficacy of NAC in reducing the incidence of CIN. While this study is not adequately powered to address this objective, analyses will be run to assess an increase in serum creatinine concentration of 25% or more from the baseline value within a 48-72 hour period after a procedure or imaging that requires the administration of contrast media as a surrogate for CIN incidence.
3. To determine NAC pharmacology administered IV or IA.

ELIGIBILITY:
Inclusion Criteria:

* Renal failure, stage 3 or worse
* Undergoing endovascular procedure with an isotonic, non ionized contrast agent
* Life expectancy at least 4 weeks from date of registration
* Platelets greater than or equal to 100,000/mm3
* Systolic pressure of greater than 90 mm Hg
* No contraindications to N-Ac or contrast agent
* Not at risk for general anesthesia

Exclusion Criteria:

* Acute renal failure
* Undergoing dialysis
* Decompensate cardiac failure
* Pregnant or nursing
* History of clinically significant reactive airway disease
* Receiving non-steroidal anti-inflammatory agent within 24 hours of study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2007-11 (Actual); Primary Completion 2014-09-15 (Actual); Study Completion 2014-09-15 (Actual)

PRIMARY OUTCOMES:
Toxicity will be graded according to NCI CTCAE version 3.0. | 2 years

SECONDARY OUTCOMES:
Baseline serum creatinine and calculated creatinine clearance to provide sample size estimates for future studies. | 2 years
To estimate the efficacy of NAC in reducing the incidence of CIN. | 2 years
To determine NAC pharmacology administered IV or IA. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Edward A Neuwelt, MD, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

REFERENCES:
- [Result] Stenstrom DA, Muldoon LL, Armijo-Medina H, Watnick S, Doolittle ND, Kaufman JA, Peterson DR, Bubalo J, Neuwelt EA. N-acetylcysteine use to prevent contrast medium-induced nephropathy: premature phase III trials. J Vasc Interv Radiol. 2008 Mar;19(3):309-18. doi: 10.1016/j.jvir.2007.11.003. PMID 18295688